CLINICAL TRIAL: NCT06287840
Title: Canadian Bone Strength Development in Children With Type 1 Diabetes Study
Brief Title: Canadian Bone Strength Development Study
Acronym: CanBSDS
Status: Recruiting | Type: Observational
Sponsor: University of Saskatchewan (Other)
Collaborators: University of Calgary (Other); The Hospital for Sick Children (Other); Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Saija Kontulainen, Professor, Associate Dean Research and Graduate Studies, Graduate Chair, University of Saskatchewan
Other Study IDs: 17-301; 488294 (Other Grant/Funding Number: Canadian Institute for Health Research)
Record Dates: First submitted 2024-02-06; First posted 2024-03-01 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Type-1 Diabetes
Keywords: Type-1 Diabetes; Bone; Growth; Children; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — Serum from Children with Type-I Diabetes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with Type-1 Diabetes: * Females: 10-11 years old
  * Males: 11-12 years old
  * Diagnosed with type-1 diabetes for at least 6 months
- Control: * Females: 10-11 years old
  * Males: 11-12 years old

SUMMARY:
The goal of this project is to learn about differences in bone development between children with and without type-1 diabetes (T1D). The main questions this study aims to answer are:

1. Assess how and when sex-specific bone developmental trajectories in the leg and arm will differ between children with T1D and control cohorts relative to the critical period of rapid skeletal growth in puberty. It is hypothesized that children with T1D will have inferior bone development, particularly lower gains in bone strength.
2. Assess why bone trajectories differ between T1D and control cohorts by identifying the role of body composition, site-specific muscle force and physical activity on differences in bone properties in female and male children with and without T1D. It is hypothesized that children with T1D will have lower gains in lean mass, muscle force, number of daily bone impacts and minutes of moderate-vigorous physical activity and will be associated with inferior gains in bone development.
3. Assess why T1D may impair sex-specific bone development by exploring the role of disease-related factors (e.g., duration, glucose control, hormones and markers of bone turnover) and fracture history on bone trajectories of children with T1D. It is hypothesized that longer exposure to T1D, poorer glucose control, alterations in hormones, lower bone formation markers and higher history of fracture will be negatively associated with bone trajectories of children with T1D.

Participant's physical growth, bone growth, muscle strength, physical activity and nutrition habits will be assessed and followed up annually for up to 4 years.

DETAILED DESCRIPTION:
The Canadian Bone Strength Development Study is a multi-site project examining differences in bone development between children with and without type-1 diabetes. Research for this study will be conducted at the University of Saskatchewan, University of Calgary, The Hospital for Sick Children (SickKids) and The Children's Hospital of Eastern Ontario (CHEO). 204 children (50% female) will be included. Participants will make 4 annual visits to the laboratory. During each laboratory visit, anthropometric measurements (e.g., height and weight), bone strength and microarchitecture, muscle strength, nutrition and physical activity will be assessed. Investigators will compare between group differences in bone growth trajectories using multilevel models.

ELIGIBILITY:
Children with Type-I Diabetes:

Inclusion Criteria

* Females: 10-11 years old.
* Males: 11 - 12 years old.
* Diagnosed with type-1 diabetes for at least 6 months.
* Capacity to give informed consent (patient and parent/guardian). Children with the capacity to give assent will do so in addition to parental consent.

Exclusion Criteria

* Consuming any medications or have additional illnesses associated with bone health, osteoporosis (including renal disease, celiac disease, hypogonadism, hyperthyroidism) or altered physical growth (precocious puberty).
* Have gone through adolescent growth spurt at study entry.

Control Group (Typically Developing Children):

Inclusion Criteria

* Females: 10-11 years old.
* Males: 11 - 12 years old.
* Capacity to give informed consent (patient and parent/guardian). Children with the capacity to give assent will do so in addition to parental consent.

Exclusion Criteria

* Have an illness or are taking medications influencing bone health or physical growth.
* Evidence of pathologic low trauma or vertebral fracture(s).
* Have gone through adolescent growth spurt at study entry.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: primary care clinic, community sample
Sampling Method: Probability Sample
Enrollment: 204 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Trabecular Thickness (μm) | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Assessed by high-resolution peripheral quantitative computed tomography (HRpQCT).
Bone Strength (Failure load) | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Assessed by high-resolution peripheral quantitative computed tomography (HRpQCT).

SECONDARY OUTCOMES:
Total, Cortical and Trabecular Bone Area (mm^2) | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Assessed by high-resolution peripheral quantitative computed tomography (HRpQCT).
Total, Cortical and Trabecular Bone Density (mg HA/cm^3) | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Assessed by high-resolution peripheral quantitative computed tomography (HRpQCT).
Cortical Thickness (μm) | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Assessed by high-resolution peripheral quantitative computed tomography (HRpQCT).
Cortical Porosity | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Assessed by high-resolution peripheral quantitative computed tomography (HRpQCT).
Trabecular Bone Volume Fraction (%) | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Assessed by high-resolution peripheral quantitative computed tomography (HRpQCT).
Trabecular Bone Number (1/mm) | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Assessed by high-resolution peripheral quantitative computed tomography (HRpQCT).
Trabecular Bone Separation (μm) | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Assessed by high-resolution peripheral quantitative computed tomography (HRpQCT).
Total Body and Hip Bone Mineral Content (g) | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Assessed by Dual-energy X-ray absorptiometry (DXA).
Total Body and Hip Areal Bone Mineral Density (g/cm^2) | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Assessed by Dual-energy X-ray absorptiometry (DXA).
Age from Peak Height Velocity (years) | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Body mass, height and sitting height will be used to estimate age from peak height velocity.
Pubertal Development | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Pubertal development will be determined using Tanner Stages (self-assessed). Participants will be asked to look at drawings of pubic hair and genital or breast development and rate what drawing best reflects their current stage of development. Each set of drawings is associated with a pubertal stage (1-5). Stage 1 indicates pre-pubertal status, stage 2-3 indicates early pubertal status, stage 4 indicates pubertal status and stage 5 indicates post-pubertal status.
Long Jump (m) | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  The furthest distance an individual can jump while starting from a standing position.
Hand Grip (N) | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  The highest amount of force one can develop by squeezing their hand. Force is measured using a hand grip dynamometer.
Bone Impacts | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Estimate of bone impact activities using a waist-worn accelerometer monitored over 7 days.
Physical Activity (minutes/day) | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Estimate of daily moderate-to-vigorous physical activity using a waist-worn accelerometer monitored over 7 days.
Food Frequency Questionnaire | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Estimate of daily intakes of calcium, protein and vitamin D. Estimates will be derived using the Food Frequency Questionnaire. Participants will be asked to recall their consumption of various foods over the last 6 months and rate their intake on a scale from Never to consuming the food item 5-6 per week. These ratings are then used to estimate the daily intake of calcum, protein and vitamin D.
Health | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  For children with type-I diabetes, investigators will record the onset of T1D (years), insulin regimen and various measures of glycemic control (e.g., HbA1c) using open-ended questionnaires and participants' medical records.
Osteocalcin | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Biochemical assessment of bone formation.
Procollagen type I N-propeptide (P1NP-N) | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Biochemical assessment of bone formation.
C-terminal telopepide (CTx) | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Biochemical assessment of bone resorption.
Sclerostin | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Biochemical assessment of bone resorption.
Insulin growth factor-1 | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Biochemical assessment of hormones.
Alkaline phosphatase | Baseline, year 1 follow-up, year 2 follow-up, year 3 follow-up
  Biochemical assessment of hormones.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada